CLINICAL TRIAL: NCT02209870
Title: The Impact of Resuscitation Quality of CPR Team by Implantation of Electronic Checklist and Alarming System Through Video-recording Analyses
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201106044RC
Record Dates: First submitted 2013-05-31; First posted 2014-08-06 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Cardiopulmonary Arrest
Keywords: Cardiopulmonary resuscitation; Teamwork; electronic checklist
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- E-checklist group: The patients after CPR team using E-checklist system
  Interventions: Behavioral: E-checklist Group

INTERVENTIONS:
Behavioral: E-checklist Group — The patient group after E-checklist system deployed

SUMMARY:
The quality of cardiopulmonary resuscitation (CPR) has been identified as an important determinants for patient survival, yet many studies revealed poor CPR guidelines compliance in real-life practice for both health care providers and lay persons. Common shortcomings identified include an insufficient number of chest compression, too rapid lung inflations, and too much hands-off time. The poor quality of CPR is associated with lower survival rate. Besides, some other problems could be found during resuscitation, such as prolonged intubation time, delayed first shock delivery or unsteady drug delivery interval. These problems can't be blamed on the only person but the teamwork. Certain measurements could improve the performance of the resuscitation team, such as audio prompt or checklist.

Methods proposed and improvised to improve the quality of CPR have included CPR assisted devices, automatic driven devices or audio prompt system. However, some of these methods are hardly incorporate with the original resuscitation process since it could be an extra workload. Therefore, the investigators try to provide an digitized checklist combined with visual and audio alarming system, which could not only minimize the workload of chart recording but also remind the team to perform essential procedures in time.

Information gained from a video-recording evaluation system had been employed to improve the resuscitation skills. The improvement of resuscitation quality also could be found through video-recording after certain intervention. It can also avoid the interference of the resuscitation and find out other harmful factors to CPR quality.

ELIGIBILITY:
Inclusion Criteria:

* Out-of-Hospital cardiac arrest patient present to NTUH ED
* Age > 18 years old
* E-checklist system applied

Exclusion Criteria:

* E-Checklist system not applied
* Video not been recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department patient Out-of-Hospital cardiac arrest patient receive CPR in NTUH Emergency Department Age > 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
return of spontaneous circulation | 60 minutes
  return of spontaneous circulation

SECONDARY OUTCOMES:
Technical skill of CPR team | 30 minutes
  including time to first shockable rhythm, no-flow time, frequency of chest compression, successful rate of rhythm conversion, Time to first shock
Non-technical skill of CPR team | 30 minutes
  Team structure and leadership, situation monitoring, workload management, communication
survival for 2 hours | 2 hours
  maintained spontaneous circulation for up to 2 hours
survival to admission | 1 day
  Survival to admission
Survival to discharge | 60 days
  Survival to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chih Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan